CLINICAL TRIAL: NCT03308773
Title: Physiology of Disease Prevention Observational Study in Clinical Practice
Brief Title: Disease Prevention in Clinical Practice Base on Patient Specific Physiology
Acronym: STOPDISEASE
Status: Enrolling by invitation | Type: Observational
Sponsor: Pacific Coast Family Medical Group (Other)
Responsible Party: Principal Investigator, John Armato, Physician, Principle investigator, Pacific Coast Family Medical Group
Other Study IDs: 2017000308
Record Dates: First submitted 2017-09-28; First posted 2017-10-13 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: PreDiabetes; Insulin Resistance; Type2 Diabetes; NASH - Nonalcoholic Steatohepatitis; Diastolic Dysfunction; Dementia; Atrial Fibrillation; Cancer; Atherosclerosis; Carotid Plaque
Keywords: Prediabetes; insulin resistance; T2DM; Carotid IMT/Plaque
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Dementia; Atrial Fibrillation; Neoplasms; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lifestyle modification in routine care of patients — Diabetes Prevention Program Lifestyle recommendations and non-investigational pharmacotherapy in routine care of patients
  Other Names: non-investigational drug in routine care of patients

SUMMARY:
It is well known that the Type 2 diabetes and vascular disease are preceded by over ten years by metabolic dysfunction and anatomic changes that can be quantified. In order to develop effective preventive strategies and reduce the cost burden to the health care system, recognition of the earliest pathophysiology of Type 2 diabetes and vascular disease is clinically relevant. The interval retrospective evaluation of data from patient records, reflect the effectiveness of the various treatments implemented in clinical practice.

Prevalence of "prediabetes" among American adults is estimated to be ~84 million, or one out of three Americans. Over a 5-7 year period approximately one third of these prediabetic individuals will progress to type 2 diabetes. Prediabetes is a heterogenous group comprised of individuals with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), and increased A1c (5.7-6.4%). Although different pathophysiologies are present in individuals with IFG and IGT, their conversion rate to overt type 2 diabetes mellitus (T2DM) is similar.

Insulin resistance is a common causal feature of many of the pathophysiologic mechanisms linking macrovascular disease and type 2 diabetes. Because hyperglycemia is the major factor responsible for the development of microvascular complications, it logically follows that prevention of progression of prediabetes to overt diabetes should retard/prevent the development of the microvascular complications. From the measurement of plasma glucose, insulin, and c-peptide levels during the oral glucose tolerance test, one can derive measures of the two core defects responsible for the development of T2DM, i.e. insulin resistance and beta cell dysfunction as well as the degree of dysglycemia.

By combining a standard medical evaluation with the evaluation of cardiovascular biomarkers, patients at intermediate risk of vascular disease can be identified. In these patients, carotid intima media thickness (IMT) and carotid plaque evaluation is offered to attempt to clarify risk.

The hypothesis of this observational study is that the characterization of the physiology and anatomy of patients at risk of developing type 2 diabetes and/or cardiovascular disease can stratify risk of developing disease and direct treatment strategies tailored to the identified physiologic defect, leading to improvements in the delay or prevention of disease.

DETAILED DESCRIPTION:
It is well known that the Type 2 diabetes and vascular disease are preceded by over ten years by metabolic dysfunction and anatomic changes that can be quantified. In order to develop effective preventive strategies and reduce the cost burden to the health care system, recognition of the earliest pathophysiology of Type 2 diabetes and vascular disease is clinically relevant. In patients with risk factors for type 2 diabetes and/or vascular disease, we have quantified this dysmetabolic state using glucose tolerance testing to quantify insulin resistance and beta cell function while measuring vascular biomarkers as well as Intima-media thickness and carotid plaque to characterize cardiovascular risk. The interval retrospective evaluation of data from patient records, reflect the effectiveness of the various treatments implemented in clinical practice.

Prevalence of "prediabetes" among American adults is estimated to be ~84 million, or one out of three Americans. Over a 5-7 year period approximately one third of these prediabetic individuals will progress to type 2 diabetes. Prediabetes is a heterogenous group comprised of individuals with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), and increased A1c (5.7-6.4%). Although different pathophysiologies are present in individuals with IFG and IGT, their conversion rate to overt type 2 diabetes mellitus (T2DM) is similar.

Prospective epidemiologic studies have demonstrated that ~40% of subjects who progress to T2DM over 5 years had Normal glucose tolerance (NGT) at baseline, suggesting that a large group of NGT subjects also are at increased T2DM risk. It has previously been demonstrated that a 1-hour plasma glucose concentration >155 mg/dl identifies a subgroup of NGT subjects with high future T2DM risk.

Further, multiple studies have demonstrated that background retinopathy, microalbuminuria, and peripheral neuropathy are present in 10-20% of prediabetic individuals. Compared with normoglycemic patients, those with prediabetes were associated with a 13-30% higher risk for composite cardiovascular disease.

Insulin resistance is a common causal feature of many of the pathophysiologic mechanisms linking macrovascular disease and type 2 diabetes. Because hyperglycemia is the major factor responsible for the development of microvascular complications, it logically follows that prevention of progression of prediabetes to overt diabetes should retard/prevent the development of the microvascular complications. From the measurement of plasma glucose, insulin, and c-peptide levels during the oral glucose tolerance test, one can derive measures of the two core defects responsible for the development of T2DM, i.e. insulin resistance and beta cell dysfunction as well as the degree of dysglycemia.

The need for improvement in the identification of asymptomatic atherosclerosis is exemplified by the observation that nearly 50% of patients suffering a first myocardial infarction have either, none or only one of the standard risk factors; smoking, diabetes, hypercholesterolemia, hypertension and family history of heart disease. By combining a standard medical evaluation with the evaluation of cardiovascular biomarkers, patients at intermediate risk of vascular disease can be identified. In these patients, carotid intima media thickness and carotid plaque evaluation is offered to attempt to clarify risk.

Further associations exist between insulin resistance and other medical conditions including; fatty liver, epicardial fat, diastolic dysfunction, arrhythmia, dementia and cancer. Quantifying insulin resistance may allow advances in preventive strategies.

Following these evaluations, a discussion of the scientific literature as well as the risk, benefits and alternatives available, a personalized treatment plan is generated. Interval reassessment is carried out as part of the routine medical care of the patients in the practice.

The hypothesis of this observational study is that the characterization of the physiology and anatomy of patients at risk of developing type 2 diabetes and/or cardiovascular disease can stratify risk of developing disease and direct treatment strategies tailored to the identified physiologic defect, leading to improvements in the delay or prevention of disease.

ELIGIBILITY:
Inclusion Criteria:

* American Diabetic Association (ADA)/American Association of Clinical Endocrinologists (AACE) criteria for patients at risk for developing type 2 diabetes

Exclusion Criteria:

* Patients with prior treatment with medications for type 2 diabetes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Internal Medicine/Endocrinology private practice in Southern California
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-01-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop type 2 diabetes based on response to oral glucose tolerance test | 6 months and an average of every 2 years through the study completion, approximately 20 years
  Patients will be monitored for up to 20 years (10 year retrospective plus 10 year prospective). The outcome measure will reflect the number of patients who develop of type 2 diabetes as evidenced by the response to oral glucose tolerance testing.
Time to development of type 2 diabetes | 6 months and an average of every 2 years through the study completion, approximately 20 years
  Patients will be monitored for up to 20 years (10 year retrospective plus 10 year prospective). The outcome measure will reflect the time to the development of type 2 diabetes as evidenced by the response to oral glucose tolerance testing.

CONTACTS AND LOCATIONS:
Overall Officials: John P Armato, MD, Principal Investigator — Providence St Josephs Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menke A, Casagrande S, Geiss L, Cowie CC. Prevalence of and Trends in Diabetes Among Adults in the United States, 1988-2012. JAMA. 2015 Sep 8;314(10):1021-9. doi: 10.1001/jama.2015.10029. PMID 26348752
- [Background] Abdul-Ghani MA, Tripathy D, DeFronzo RA. Contributions of beta-cell dysfunction and insulin resistance to the pathogenesis of impaired glucose tolerance and impaired fasting glucose. Diabetes Care. 2006 May;29(5):1130-9. doi: 10.2337/diacare.2951130. PMID 16644654
- [Background] Abdul-Ghani MA, Jenkinson CP, Richardson DK, Tripathy D, DeFronzo RA. Insulin secretion and action in subjects with impaired fasting glucose and impaired glucose tolerance: results from the Veterans Administration Genetic Epidemiology Study. Diabetes. 2006 May;55(5):1430-5. doi: 10.2337/db05-1200. PMID 16644701
- [Background] Diabetes Prevention Program Research Group. The prevalence of retinopathy in impaired glucose tolerance and recent-onset diabetes in the Diabetes Prevention Program. Diabet Med. 2007 Feb;24(2):137-44. doi: 10.1111/j.1464-5491.2007.02043.x. PMID 17257275
- [Background] DREAM Trial Investigators; Dagenais GR, Gerstein HC, Holman R, Budaj A, Escalante A, Hedner T, Keltai M, Lonn E, McFarlane S, McQueen M, Teo K, Sheridan P, Bosch J, Pogue J, Yusuf S. Effects of ramipril and rosiglitazone on cardiovascular and renal outcomes in people with impaired glucose tolerance or impaired fasting glucose: results of the Diabetes REduction Assessment with ramipril and rosiglitazone Medication (DREAM) trial. Diabetes Care. 2008 May;31(5):1007-14. doi: 10.2337/dc07-1868. Epub 2008 Feb 11. PMID 18268075
- [Background] Asghar O, Petropoulos IN, Alam U, Jones W, Jeziorska M, Marshall A, Ponirakis G, Fadavi H, Boulton AJ, Tavakoli M, Malik RA. Corneal confocal microscopy detects neuropathy in subjects with impaired glucose tolerance. Diabetes Care. 2014 Sep;37(9):2643-6. doi: 10.2337/dc14-0279. Epub 2014 Jun 26. PMID 24969581
- [Background] Gibbons CH, Goebel-Fabbri A. Microvascular Complications Associated With Rapid Improvements in Glycemic Control in Diabetes. Curr Diab Rep. 2017 Jul;17(7):48. doi: 10.1007/s11892-017-0880-5. PMID 28526993
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Armato J, DeFronzo RA, Abdul-Ghani M, Ruby R. Successful treatment of prediabetes in clinical practice: targeting insulin resistance and beta-cell dysfunction. Endocr Pract. 2012 May-Jun;18(3):342-50. doi: 10.4158/EP11194.OR. PMID 22068250
- [Background] Huang Y, Cai X, Mai W, Li M, Hu Y. Association between prediabetes and risk of cardiovascular disease and all cause mortality: systematic review and meta-analysis. BMJ. 2016 Nov 23;355:i5953. doi: 10.1136/bmj.i5953. PMID 27881363
- [Derived] Armato JP, DeFronzo RA, Abdul-Ghani M, Ruby RJ. Successful treatment of prediabetes in clinical practice using physiological assessment (STOP DIABETES). Lancet Diabetes Endocrinol. 2018 Oct;6(10):781-789. doi: 10.1016/S2213-8587(18)30234-1. Epub 2018 Sep 14. PMID 30224284